CLINICAL TRIAL: NCT02727465
Title: Host-pathogen Interactions in Meningococcal Disease: Finding the Key That Fits the Lock
Acronym: Lock and Key
Status: Withdrawn | Type: Observational
Sponsor: Public Health England (Other Government)
Responsible Party: Sponsor
Other Study IDs: Lock and Key
Record Dates: First submitted 2016-03-09; First posted 2016-04-04 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Meningitis
MeSH Terms: conditions — Meningitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — DNA of bacteria and cases
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- meningitis cases: any individual with culture-confirmed IMD in England from 01 September 2015 to 31 August 2019 with written informed consent from the individual, the parent (for children aged <16 years) or next-of-kin (for non-survivors)
  Interventions: Other: Meningitis cases

INTERVENTIONS:
Other: Meningitis cases — None - blood draw only

SUMMARY:
At any time, around 10% of people carry meningococcal bacteria in the nose and throat, which can cause meningitis, blood poisoning and other serious illnesses. Most people carry these bacteria and never become ill, yet a very small proportion go on to develop these illnesses which can result in life long disabilities or death. The mechanism by which this happens is poorly understood and has been studied in various ways, usually focussing on the bacteria or on the individual, but none has given a definitive answer. This study will be the first of its kind and will assess the interaction between the host and the bacteria at the genetic level, through genetic mapping, helping us to understand what makes some people susceptible to this infection.

DETAILED DESCRIPTION:
At any time, around 10% of people carry meningococcal bacteria in the nose and throat, which can cause meningitis, blood poisoning and other serious illnesses. Most people carry these bacteria and never become ill, yet a very small proportion go on to develop these illnesses which can result in life long disabilities or death. The mechanism by which this happens is poorly understood and has been studied in various ways, usually focussing on the bacteria or on the individual, but none has given a definitive answer. This study will be the first of its kind and will assess the interaction between the host and the bacteria at the genetic level, through genetic mapping, helping us to understand what makes some people susceptible to this infection.

ELIGIBILITY:
Inclusion Criteria:

* any individual with culture-confirmed IMD in England from 01 September 2015 to 31 August 2019
* written informed consent from the individual, the parent (for children aged <16 years) or next-of-kin (for non-survivors)

Exclusion Criteria:

* any individual who does not fulfil the inclusion criteria

Temporary Exclusion Criteria:

* Critically-ill patients and/or their family member will be only approached when the patient starts recovering from their illness or after they are deceased, on the advice of their clinical team.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: any individual with culture-confirmed IMD in England from 01 September 2015 to 31 August 2019 with written informed consent from the individual, the parent (for children aged <16 years) or next-of-kin (for non-survivors)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
informed consent obtained for all culture-confirmed IMD to sequence their genome. | up to 55 months
  enrol cases

SECONDARY OUTCOMES:
creation of a functional database linking anonymised whole genome human and meningococcal sequences with data collected through national surveillance | up to 55 months
  construction of reference database
detailed genetic analysis on human-pathogen pairs, focussing particularly on (but not restricted to) the human complement system and the respective meningococcal binding proteins. | up to 55 months
  Genetic analysis
visualising potential host-pathogen interactions through computer modelling | up to 55 months
  computer modelling

CONTACTS AND LOCATIONS:
Overall Officials: Shamez Ladhani, MD PhD, Principal Investigator — Public Health England
Locations (1):
- All NHS hospitals, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No